CLINICAL TRIAL: NCT03458975
Title: Targeted Delivery of Chemotherapy With Ultrasound and Microbubbles
Brief Title: Targeted Delivery of Chemotherapy With Ultrasound and Microbublles
Acronym: SONCHIMIO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRTK15-TL/SONCHIMIO
Record Dates: First submitted 2018-03-02; First posted 2018-03-08 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Cancer; Hepatic Metastases
Keywords: microbubbles; sonoporation; hepatic metastases of colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Selected liver metastases of the patient (Active Comparator): Liver metastases randomized to receive sonoporation (US waves + gaseous microbubbles). The patient continue to receive the usual systemic chemotherapy
  Interventions: Radiation: MRI; Radiation: Perfusion CT scan; Other: Contrast enhanced ultrasound; Drug: Sonoporation
- Not-selected liver metastases of the patient (Placebo Comparator): Liver metatstases not randomized to receive sonoporation (US waves + gaseous microbubbles). The patient continue to receive the usual systemic chemotherapy like the active comparator arm
  Interventions: Radiation: MRI; Radiation: Perfusion CT scan; Other: Contrast enhanced ultrasound

INTERVENTIONS:
Radiation: MRI — Magnetic Resonance Imaging
Radiation: Perfusion CT scan — Perfusion Computerized tomography scan
Other: Contrast enhanced ultrasound — Contrast enhanced ultrasound
Drug: Sonoporation — Gaseous microbubbles (Sonovue) combinated with Ultrasounds
  Arms: Selected liver metastases of the patient

SUMMARY:
The oscillations of ultrasound (US) contrast agent microbubbles under their activation by US waves engender a modulation of the permeability of biological barriers amplifying hence the extravasation of drugs and/or fluorescent markers through a process known as sonoporation. In such a way, the bioavailability of the therapeutic agent is augmented only in the area where US waves are focused. The objective now is to translate this therapeutic approach to the clinic by performing a feasibility study with the development of a therapy regime optimized for hepatic metastases of colorectal cancer.

In order to demonstrate the clinical feasibility of the therapeutic approach based on ultrasound and microbubbles, we will focus on patients with liver metastases of colorectal cancer treated with monoclonal antibodies in combination with chemotherapy.

DETAILED DESCRIPTION:
Despite the increasing number of active molecules and the availability of news targeted therapies for cancer, therapeutic achievements remain modest for a number of tumor types. One of the major obstacles is inherent to the absence of specific delivery in the tumor tissue.

We have demonstrated recently that the oscillations of ultrasound (US) contrast agent microbubbles under their activation by US waves engender a modulation of the permeability of biological barriers amplifying hence the extravasation of drugs and/or fluorescent markers through a process known as sonoporation. In such a way, the bioavailability of the therapeutic agent is augmented only in the area where US waves are focused. The objective now is to translate this therapeutic approach to the clinic by performing a feasibility study with the development of a therapy regime optimized for hepatic metastases of colorectal cancer.

In order to demonstrate the clinical feasibility of the therapeutic approach based on ultrasound and microbubbles, we will focus on patients with liver metastases of colorectal cancer treated with monoclonal antibodies in combination with chemotherapy.

The work aims into evaluating the therapeutic efficacy of the proposed approach on a number of selected patients. We will follow the usual treatment schemes and we will apply imaging protocols to visualize tumor progression.

This technique of optimization of the intratumoral availability of anticancer drugs and based on sonoporation will improve the efficacy and safety of systemic chemotherapy by providing increased tumor uptake relative to normal tissue. This technique provides an ideal and easy strategy to optimize intratumoral drug delivery.

ELIGIBILITY:
Inclusion Criteria:

* patient with liver metastases from colorectal cancer; patient with minimum two liver metastases which satisfy all the following criteria: diameter between 10 and 35 mm; arterially enhancing liver metastases detected with contrast enhanced ultrasound (CEUS); measurable liver metastases with CT-scan (Acceptability of a patient with more than 4 metastases or a patient with an odd number of metastases ≥ 2).
* age ≥ 18 years;
* ECOG/OMS 0-1;
* life expectancy of at least 12 weeks;
* adequate bone marrow, liver and kidney function;
* written informed consent obtained from subject;
* subjects covered by or having the rights to social security;
* bi-weekly chemotherapy regimen
* neo-adjuvant standard chemotherapy or palliative standard chemotherapy (first or second metastatic line) following the recommendations in force (national thesaurus of digestive oncology - colorectal cancer chapter: Phelip JM, Benhaim L, Bouché O, Christou N, Desolneux G, Dupré A, Léonard D, Michel P, Penna C, Rousseaux B, Tougeron D, Tournigand C. "Cancer colorectal métastatique". Thésaurus National de Cancérologie Digestive, Janvier 2019, http://www.tncd.org).

Exclusion Criteria:

* Previous local treatment of selected liver metastases (radiofrequency, radioembolization, …);
* Indication for local ablative therapy of selected liver metastasis (radiofrequency ablation or other validated hepatic-directed modality of treatment);
* Previous malignancy other than colorectal adenocarcinoma within 3 years prior to the inclusion with the exception for curatively treated basal cell carcinoma of the skin and/or curatively resected in situ cervical or breast cancer;
* Known contraindication to the injection of Sonovue®, of Gadolinium, of iodated contrast agent;
* contraindication to MRI or perfusion CT scan;
* Patient under legal protection;
* Pregnant or lactating woman, or woman with ability to procreate and without contraception;
* Inclusion in another therapeutic trial
* Uracilemia greater than or equal to 150ng/mL (suggestive of a complete DPD deficiency).
* Presence of any material with potential interaction with ultrasound beam (metal, etc.) or healing tissue, and which cannot be bypassed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Objective response for liver metastases | 2 months
  Objective response for liver metastases with spiral CT scan and defined as decrease of at least 30% in the longer diameter of each selected liver metastases

SECONDARY OUTCOMES:
Safety | Day 3, Day 17, Day 32, Day 47
  Safety based on National Cancer Institute (NCI), Common Terminology Criteria for Adverse events (CTCAE)
Tolerance | Day 3, Day 17, Day 32, Day 47
  Tolerance based on National Cancer Institute (NCI), Common Terminology Criteria for Adverse events (CTCAE)
Maximum percent reduction in tumor density on CT scan | 2 months
  Maximum percent reduction in tumor density (Hounsfield units) from baseline
Maximum percent reduction in tumor density on MRI | 2 months
  Maximum percent reduction in tumor density from baseline
Assessment of tumor vascularity by Perfusion CT scan | 2 months
  Assessment of tumor vascularity with Perfusion CT scan
Assessment of tumor vascularity by MRI | 2 months
  Assessment of tumor vascularity with MRI
Assessment of tumor vascularity by Dynamic Contrast-Enhanced US (DCE-US) | 2 months
  Assessment of tumor vascularity with Dynamic Contrast-Enhanced US (DCE-US)
Dosage of antibody anti-VEGF or anti-EGFR | Day1, Day 3, Day 15, Day 17, Day 32, Day 45
  Measures of serum concentration of antibody anti-VEGF or anti-EGFR
Dosage of antibody anti-VEGF or anti-EGFR by ELISA test | Day1, Day 3, Day 15, Day 17, Day 32, Day 45
  Pharmacokinetic of antibody anti-VEGF or anti-EGFR
Dosage of cytokines | Day1, Day 3, Day 15, Day 17, Day 32, Day 45
  Dosage of cytokines

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Hépatogastro-entérologie CHRU de TOURS, Tours, France

IPD SHARING:
Plan to Share IPD: No